CLINICAL TRIAL: NCT04155892
Title: A Prospective Observational Study Evaluating Extubation Criteria in Children Less Than 8 Years of Age With Upper Respiratory Infection Undergoing Outpatient or Day Hospital Based Surgery
Brief Title: Evaluation of Extubation Criteria in Children With Upper Respiratory Infection (URI)
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00056059
Record Dates: First submitted 2019-11-05; First posted 2019-11-07 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-10

CONDITIONS: Upper Respiratory Tract Infections
Keywords: Extubation criteria; Pediatric Anesthesia; Outpatient surgery
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- URI group: This group includes participants <8 years of age undergoing elective procedures with a score of at least 3 on our pre-operative URI survey.
- non-URI group: This group includes participants <8 years of age undergoing elective procedures with no URI symptoms or recent URI.

SUMMARY:
The investigators are currently completing a data collection to try to optimize pediatric patients' preoperative screening, in the setting of an upper respiratory infection.

DETAILED DESCRIPTION:
The objectives of this study are to evaluate various extubation criteria and their predictive value for successful extubation in non-cardiac surgical procedures. To evaluate the predictive value of room air oxygen and an original preoperative URI questionnaire in pediatric patients with URI or URI symptoms.

ELIGIBILITY:
Inclusion Criteria:

* All study participants must be undergoing general anesthesia and surgery with an endotracheal tube
* The URI group will be participants with a score of at least 3 on our pre-operative URI survey, with planned airway instrumentation with an endotracheal tube (ETT) for their surgical procedure who are to be discharged same day or on postoperative day 1.
* The non URI group will be participants undergoing elective procedures with no URI symptom or recent URI. Defined as no URI or "allergy" symptom within the past 6 weeks and a score of 1 or less on the URI survey, with planned airway instrumentation with an ETT for their surgical procedure who are to be discharged same day or on postoperative day 1.

Exclusion Criteria:

* History of home oxygen use or ventilator dependence,
* Patients undergoing emergent procedures.
* Patients with cyanotic congenital heart disease.
* Patients receiving a surgical procedure where the duration of post procedure
* admission is anticipated to be greater or equal to 2 postoperative days.
* Patients undergoing anesthesia for imaging procedures alone.
* Patients who are extubated deep intentionally.
* Patients intended to be managed with supraglottic airway.
* Patients undergoing total IV anaesthesia (TIVA).

Max Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: * All study participants must be < 8 years of age and undergoing general anesthesia and surgery with an endotracheal tube
  * The URI group will be participants with a score of at least 3 on our pre-operative URI survey, with planned airway instrumentation with an ETT for their surgical procedure who are to be discharged same day or on postoperative day 1.
  * The non URI group will be participants undergoing elective procedures with no URI symptom or recent URI. Defined as no URI or "allergy" symptom within the past 6 weeks and a score of 1 or less on the URI survey, with planned airway instrumentation with an ETT for their surgical procedure who are to be discharged same day or on postoperative day 1.
Sampling Method: Non-Probability Sample
Enrollment: 760 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-03 (Actual)

PRIMARY OUTCOMES:
The rate of successful extubation in children with at least 3 of the five criteria present | Day 1
  The 5 criteria (facial grimace, eye opening, conjugate gaze, purposeful movement, and tidal volume > 5 cc/kg)
Rate of participants with an extubation requiring intervention | Day 1
  The quality of extubation will be graded as successful, intervention required or major intervention required
Rate of participants with an extubation requiring major intervention | Day 1
  The quality of extubation will be graded as successful, intervention required or major intervention required
Rate of participants with a successful extubation | Day 1
  The quality of extubation will be graded as successful, intervention required or major intervention required

SECONDARY OUTCOMES:
Rate of on time and anticipated discharge from the hospital | Up to 5 days after discharge
Rate of patients seeking additional care following discharge for respiratory related symptoms | Up to 5 days after discharge
Preoperative room air oxygen saturation | Day 1
Rate of extubation success per the number of factors present at time of extubation | Day 1
  Rate of success at the presence of 3 to 6 predictors (eye opening, facial grimace, purposeful movement, conjugate gaze, tidal volume > 5 cc/kg, and ETCO2<56 mmHg) at time of extubation

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Templeton, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No